CLINICAL TRIAL: NCT02317354
Title: Patient Expectations When Enrolling in a Phase I/II RS1 Ocular Gene Transfer Clinical Trial
Brief Title: People s Expectations When Enrolling in a Phase I/II RS1 Ocular Gene Transfer Clinical Trial
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150041; 15-EI-0041
Record Dates: First submitted 2014-12-13; First posted 2014-12-16 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-11-20

CONDITIONS: Retinoschisis; X-Linked
Keywords: X-Linked; Retinoschisis
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

-X-linked retinoschisis (XLRS) is an inherited eye condition. Researchers want to learn more about how people with XLRS choose to take part in research studies. They hope to find ways to help other people make decisions about joining early phase trials

Objective:

-To learn more about how people think and feel about taking part in early phase research.

Eligibility:

-Adults age 18 or older with diagnosed XLRS. They must be eligible to be screened for a Phase I/II ocular gene transfer clinical trial.

Design:

* Participants will be screened for the XLRS gene transfer study. They will be interviewed:
* Eligible participants who join the study - before the gene transfer procedure, then 3 months and 12 months after it.
* Eligible participants who do not join the study - after their screening visit and 3 months and 12 months later.

<TAB>- Participants who are screened but ineligible - after their screening visit.

<TAB>- Participants who choose not to be screened - at the time they make the decision and 1 year later.

* Interviews will ask for the participants thoughts about the clinical trial and why they chose to take part or not. The interviews will be recorded.
* On the day of interview 1, participants will fill out a survey about their mood and personality.
* On the days of interviews 2 and 3, participants will fill out a survey about their mood.
* Interviews may be done in person or by phone. Surveys can be done online or through the mail. Or they can be done in person at the NIH Clinical Center.

DETAILED DESCRIPTION:
Objective: The objective of this study is to understand the factors that influence patient expectations when enrolling in an early-phase RS1 ocular gene transfer clinical trial and to assess the psychological impact of patient expectations over time.

Study Population: Up to 50 adults with X-linked retinoschisis who are eligible to be screened for a Phase I/II ocular gene transfer clinical trial will be included in this study. We hope to capture the experience of those actively engaged in the decision-making process who may choose not to participate in the clinical trial or who may receive gene transfer.

Design: This is a prospective qualitative interview study with quantitative questionnaires. Participation will involve up to three interviews with questionnaires over one year. Interviews may take place in person at the National Institutes of Health Clinical Center (NIH CC) or by telephone and will focus on how the interviewee came to the decision to participate (not to participate) in the early-phase ocular gene transfer trial. Interviews will be transcribed verbatim, coded by two independent coders, and analyzed thematically. Participants will also be asked to complete a questionnaire that measures dispositional optimism, resilience, and general mood states using instruments that have been shown to be valid and reliable in both the general population and in clinical samples. Information collected from these surveys will supplement information collected during the qualitative interview and will provide information about constructs that are difficult to assess during a brief interview.

Outcome Measures: The primary outcomes of this study include a description of what research participants expect when choosing to enroll in an early-phase clinical trial and a description of the psychological impact, over time, of having high expectations

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants may be eligible to take part in this study if they:

* Are 18 years of age or older.
* Have a molecular diagnosis of XLRS and are eligible to be screened for a Phase I/II ocular gene transfer clinical trial.
* Are able to understand and comply with the procedures of this study.

EXCLUSION CRITERIA:

Participants may not be able to take part in this study if they:

* Have eye findings or other medical conditions that would preclude consideration for participation in a Phase I/II ocular gene transfer clinical trial.
* Are receiving experimental treatment for XLRS in another research study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12-13; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Desc. expectation pt enroll ct | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Turriff, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jansen LA. Two concepts of therapeutic optimism. J Med Ethics. 2011 Sep;37(9):563-6. doi: 10.1136/jme.2010.038943. Epub 2011 May 7. PMID 21551464
- [Background] Appelbaum PS, Roth LH, Lidz C. The therapeutic misconception: informed consent in psychiatric research. Int J Law Psychiatry. 1982;5(3-4):319-29. doi: 10.1016/0160-2527(82)90026-7. No abstract available. PMID 6135666